CLINICAL TRIAL: NCT01669018
Title: The Supra Sacral Parallel Shift (SSPS) - Ultrasound Guided Blockade of the Lumbar Plexus
Brief Title: Ultrasound Guided Blockade of the Lumbar Plexus - the Supra Sacral Parallel Shift
Acronym: SSPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Thomas F. Bendtsen, Consultant anesthetist, associate professor, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SSPS-1-10-72-366-12
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumbar ultrasound trident (LUT) (Active Comparator): Lumbar plexus block using LUT technique
  Interventions: Procedure: Lumbar plexus block using LUT technique
- Supra Sacral Parallel Shift (SSPS) (Experimental): Lumbar plexus block using SSPS technique
  Interventions: Procedure: Lumbar plexus block using SSPS technique

INTERVENTIONS:
Procedure: Lumbar plexus block using LUT technique — Lumbar plexus block guided by ultrasound and nerve stimulation with the patient in the lateral position and the probe in the parasagittal plane inserting the block needle between the transverse processes of L3 and L4 until an appropriate neuromuscular response is produced.
  Arms: Lumbar ultrasound trident (LUT)
Procedure: Lumbar plexus block using SSPS technique — Lumbar plexus block guided by ultrasound and loss of resistance (LOR) with the patient in the lateral position and the probe in the parasagittal plane inserting the block needle between the transverse process of L5 and the sacral bone until an appropriate LOR is produced.
  Arms: Supra Sacral Parallel Shift (SSPS)

SUMMARY:
Anesthesia for hip surgery can be performed with ultrasound guided blockade of the mesh of nerves (the lumbar plexus) supplying the hip region from the lumbar spinal nerves. This is a relevant technique in patients with severe cardiac comorbidity. The technique is a safer alternative compared to general or spinal anesthesia in these fragile patients.

The most recognized technique with ultrasound guidance (Karmakars technique) is technically demanding and based on injection of local anesthetic relatively close to the exit of the spinal nerves from the spine. The risk is spread of local anesthetic to the spinal canal prompting a risk of low blood pressure. This may be fatal in high risk patients.

The investigators have developed a simple technique based on injection away from the spinal canal. The investigators expect minimal risk of spread of local anesthetic to the spinal canal with this technique.

This randomized, double blinded trial compares the new technique to the established technique of ultrasound guided blockade of the lumbar plexus.

The hypothesis is that the new technique has a higher success rate with reduced effect on blood pressure for ultrasound guided lumbar plexus block compared to the established technique.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* ASA I (American Society of Anesthesiologists physical status classification)

Exclusion Criteria:

* volunteers who are not able to cooperate
* volunteers who do not understand and speak danish
* daily use of analgesics
* allergy to local analgesics or contrast agents
* abuse of medicine or alcohol
* volunteers with technical impediments of the planned interventions

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Success of complete sensory blockade of dermatomes L2, L3, L4, L5, S1 | 30 minutes after injection of local anesthetic

SECONDARY OUTCOMES:
Plasma lidocaine level (mcg/mL) | 0, 5, 10, 20, 40, 60, and 90 minutes after injection of local anesthetic
  Chromatography analysis
Block performance time | From start of probe on the skin until injection of local anesthetic is completed
Patient satisfaction | Immediately after completion of injection of local anesthetic
Mean arterial blood pressure (MAP) | 5 minutes after completion of injection of local anesthetic
  Absolute measure and relative change from pre-block measure
Cost-effectiveness | Block performance time period
  Estimated as incremental cost-effectiveness ratio
Sensory blockade of each dermatome L1, L2, L3, L4, L5, S1, S2, and S3 (cold, warmth, touch, pain) | 30 minutes after completed injection of local anesthetic
Sensory blockade of the femoral nerve (cold, warmth, touch, pain) | 30 minutes after completion of injection of local anesthetic
Motor blockade of the femoral nerve | 40 minutes after completion of injection of the local anesthetic
Motor blockade of the obturator nerve | 40 minutes after completion of injection of the local anesthetic
Perineural spread of local anesthetic (with contrast) estimated with MRI | 60 minutes after completion of injection of local anesthetic

CONTACTS AND LOCATIONS:
Overall Officials: Else Tønnesen, Professor, Study Chair — Faculty of Health, Aarhus University
Locations (1):
- Department of Anesthesiology, Aarhus University Hospital, Aarhus, Denmark